CLINICAL TRIAL: NCT00453882
Title: An Evaluation of Ureteral Flow After Temporary Bilateral Uterine Artery Occlusion During Conservative Gynecological Procedures
Brief Title: Uretal Flow Assessment During Gynecological Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 300-06-003
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Conservative Gynecological Procedures
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: flostat (TM) System

SUMMARY:
The objective is to evaluate the feasibility of using color Doppler ultrasound in ureteral flow assessment after uterine artery occlusion during a conservative gynecological procedure.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for conservative gynecological procedure
* At least 25 years of age
* Cervix suitable for tenaculum placement
* Provides written informed consent.

Exclusion Criteria:

* Pregnancy
* One or more lower uterine segment fibroids
* Hydronephrosis as determined by renal ultrasound pre-procedurally
* Clinical diagnosis of urinary tract infection (UTI)
* In the medical judgment of the physician, such a procedure may compromise the patient's condition
* Inability to achieve bilateral occlusion with the clamp placement during the procedure.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Ability to evaluate ureteric jets
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: David Robinson, MD, Study Director — Ethicon, Inc.
Locations (1):
- Holy Cross Medical Group, Fort Lauderdale, Florida, United States